CLINICAL TRIAL: NCT00536237
Title: Part A: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Effects of MK0524 Compared to Placebo Part B: A Dose-Ranging Study to Evaluate the Tolerability of MK0524 and Its Effects on Niacin-Induced Flushing in Lipid Clinic Patients
Brief Title: MK0524A Phase IIb Study (0524A-011)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-011; MK0524A-011; 2007_618
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Flushing
MeSH Terms: conditions — Flushing | interventions — Duration of Therapy; Niacin; MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Comparator: niacin / Duration of Treatment: 17 Weeks
Drug: MK0524A, niacin (+) laropiprant / Duration of Treatment: 17 Weeks
Drug: Comparator: placebo (unspecified) / Duration of Treatment: 17 Weeks

SUMMARY:
Part A: This study will determine that MK0524 is well tolerated and does not effect lipids and blood glucose when given alone.

Part B: Determine dose ranges for MK0524 and MK0524 plus Niaspan(R) on the effects of lipids and blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 to 70 years of age for whom treatment with Niacin would be appropriate but who are not taking > 50mg at screening
* Must be willing to complete electronic diary

Exclusion Criteria:

* Subject is having menopausal hot flashes and/or receiving hormone replacement therapy (HRT)
* You have a history of cancer, gout, peptic ulcers, diabetes, liver, heart disease or high blood pressure or you are HIV positive
* You consume more than 14 alcoholic drinks per week or more than 2 drinks per day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2004-08; Primary Completion 2005-02 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To determine the effect of MK0524A on lipids and blood glucose | 17 Weeks

SECONDARY OUTCOMES:
To establish the dose for limiting flushing symptoms induced by NIASPAN (R) | 17 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Paolini JF, Mitchel YB, Reyes R, Kher U, Lai E, Watson DJ, Norquist JM, Meehan AG, Bays HE, Davidson M, Ballantyne CM. Effects of laropiprant on nicotinic acid-induced flushing in patients with dyslipidemia. Am J Cardiol. 2008 Mar 1;101(5):625-30. doi: 10.1016/j.amjcard.2007.10.023. Epub 2007 Dec 21. PMID 18308010